CLINICAL TRIAL: NCT02383862
Title: Incorporating PROMIS Symptom Measures Into Primary Care Practice
Brief Title: PROMIS Measures in Primary Care Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kurt Kroenke, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1410447721
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Sleep; Pain; Anxiety; Depression; Fatigue
Keywords: Sleep; Pain; Anxiety; Depression; Fatigue; PROMIS; primary care
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Feedback Group (Experimental): Patients whose clinician received baseline PROMIS symptom scores at the time of their clinic visit
  Interventions: Other: Feedback Group
- Control Group (No Intervention): Patients whose clinician did not receive baseline PROMIS symptom scores at the time of their clinic visit

INTERVENTIONS:
Other: Feedback Group — The intervention will consist of feedback provided to clinicians in the form of patients' baseline PROMIS scores
  Arms: Feedback Group

SUMMARY:
The purpose of this study is to determine the effectiveness of providing PROMIS Profile Scale scores (e.g., sleep, pain, anxiety, depression, energy/fatigue) to physicians on patients' symptoms.

DETAILED DESCRIPTION:
The SPADE symptoms (sleep, pain, anxiety, depression, and energy/fatigue) are the most common yet undertreated symptoms in clinical practice. Using the PROMIS (Patient-Reported Outcome Measurement Information System) Profile Scales as a measure of SPADE symptoms, this study will determine the effectiveness of providing patient symptom scores to clinicians, identify barriers and facilitators to the clinical use of such scores, and evaluate the psychometric properties of the PROMIS Profile Scales in a primary care population.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Adults ≥ 18 years of age,
* Receiving care from a participating primary care physician
* Report a moderate level of severity ( ≥ 4 on a 0 to 10 scale) on at least one of 5 symptoms (sleep, pain, anxiety, depression, energy/fatigue) based on a 5-item screener.

Physicians

* Primary care physicians within the Indiana University Health and Eskenazi Health systems

Exclusion Criteria:

Patients

* Patients less than 18 years of age
* Patients who do not receive care from a participating primary care physician
* Patients who have less than a moderate level of severity (less than 4 on a 0 to 10 item scale) on each of the 5 symptoms (sleep, pain, anxiety, depression, energy/fatigue) based on a 5-item screener.

Physicians:

* Primary care physicians who do not practice within the Indiana University Health or Eskenazi Health systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Kroenke, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Kroenke K, Stump TE, Kean J, Talib TL, Haggstrom DA, Monahan PO. PROMIS 4-item measures and numeric rating scales efficiently assess SPADE symptoms compared with legacy measures. J Clin Epidemiol. 2019 Nov;115:116-124. doi: 10.1016/j.jclinepi.2019.06.018. Epub 2019 Jul 19. PMID 31330252
- [Derived] Talib TL, DeChant P, Kean J, Monahan PO, Haggstrom DA, Stout ME, Kroenke K. A qualitative study of patients' perceptions of the utility of patient-reported outcome measures of symptoms in primary care clinics. Qual Life Res. 2018 Dec;27(12):3157-3166. doi: 10.1007/s11136-018-1968-3. Epub 2018 Aug 14. PMID 30109471
- [Derived] Kroenke K, Talib TL, Stump TE, Kean J, Haggstrom DA, DeChant P, Lake KR, Stout M, Monahan PO. Incorporating PROMIS Symptom Measures into Primary Care Practice-a Randomized Clinical Trial. J Gen Intern Med. 2018 Aug;33(8):1245-1252. doi: 10.1007/s11606-018-4391-0. Epub 2018 Apr 5. PMID 29623512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between March 2015 and April 2016 in primary care outpatient clinics.
Pre-assignment Details: In clinic, patients who had 1≤ SPADE (sleep, pain, anxiety, depression low energy/fatigue) symptoms, consented and provided authorization, completed PROMIS (Patient-Reported Outcome Measurement Information System), and then were randomized to a feedback or control group. Patients unable to complete enrollment prior to the encounter were excluded.
Period: Baseline
Arm/Group | Feedback Group | Control Group
Started | 151 | 149
Completed | 151 | 149
Not Completed | 0 | 0
Period: 3 Month Follow up
Arm/Group | Feedback Group | Control Group
Started | 151 | 149
Completed | 128 | 128
Not Completed | 23 | 21
Not completed — Lost to Follow-up | 23 | 21

BASELINE CHARACTERISTICS:
Population: Patients with 1 or more SPADE symptoms who completed enrollment (e.g., consent, authorization, baseline questionnaire, randomization)
Groups:
- Total: Total of all reporting groups
Arm/Group | Feedback Group | Control Group | Total
Number analyzed (Participants) | 151 | 149 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (14.1) | 48.2 (14.7) | 49.4 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 104 | 215
  Male | 40 | 45 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 123 | 120 | 243
  Unknown or Not Reported | 23 | 22 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 79 | 69 | 148
  White | 65 | 70 | 135
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 2 | 5 | 7
PROMIS Composite T-score [Mean (Standard Deviation); unit: T-score] — The 20-item PROMIS questionnaire (composed of 4-item scales for each of the 5 SPADE symptoms) assesses the extent to which patients experience problems with SPADE symptoms over the past 7 days using a 5-point Likert scale. Each PROMIS scale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. The composite PROMIS T-score is the sum of the 5 symptom T-scores divided by 5. Higher scores reflect greater symptom severity.
  T-score | 58.3 (7.6) | 58.4 (6.4) | 58.3 (7.0)
PROMIS Sleep T-score [Mean (Standard Deviation); unit: T-score] — The 4-item PROMIS subscale for sleep assesses the extent to which patients experience problems with sleep over the past 7 days using a 5-point Likert scale. The sleep subscale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. Higher scores reflect more severe sleep problems.
  T-score | 58.3 (9.4) | 58.1 (8.7) | 58.2 (9.0)
PROMIS Pain T-score [Mean (Standard Deviation); unit: T-score] — The 4-item PROMIS subscale for pain assesses the extent to which patients experience problems with pain over the past 7 days using a 5-point Likert scale. The pain subscale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. Higher scores reflect greater pain.
  T-score | 61.5 (9.3) | 61.4 (9.5) | 61.5 (9.4)
PROMIS Anxiety T-score [Mean (Standard Deviation); unit: T-score] — The 4-item PROMIS subscale for anxiety assesses the extent to which patients experience anxiety symptoms over the past 7 days using a 5-point Likert scale. The anxiety subscale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. Higher scores reflect greater anxiety.
  T-score | 59.0 (10.1) | 59.2 (8.7) | 59.1 (9.4)
PROMIS Depression T-score [Mean (Standard Deviation); unit: T-score] — The 4-item PROMIS subscale for depression assesses the extent to which patients experience depressive symptoms over the past 7 days using a 5-point Likert scale. The depression subscale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. Higher scores reflect greater depression.
  T-score | 55.8 (10.4) | 56.0 (9.1) | 55.9 (9.8)
PROMIS Fatigue T-score [Mean (Standard Deviation); unit: T-score] — The 4-item PROMIS subscale for fatigue assesses the extent to which patients experience problems with fatigue over the past 7 days using a 5-point Likert scale. The fatigue subscale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. Higher scores reflect greater fatigue.
  T-score | 56.8 (10.1) | 57.2 (9.9) | 57.0 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PROMIS Composite T-Score at 3-Month Follow-up
Description: The 20-item PROMIS questionnaire (composed of 4-item scales for each of the 5 SPADE symptoms) was administered to participants at baseline and at 3 month follow up. PROMIS assesses the extent to which patients experience problems with SPADE symptoms over the past 7 days using a 5-point Likert scale. Higher scores reflect greater symptom severity. To assess the effects of feedback on SPADE symptom improvement, group differences in the change in PROMIS composite T-scores from baseline to 3 month follow up (baseline PROMIS T-score - 3 month PROMIS T-score) were calculated. Positive change scores are indicative of symptom improvement.
Time Frame: baseline and 3 month follow up
Population: Multiple imputation was used to determine follow-up scores for nonrespondents.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 151 | 149
T-score | 3.48 (0.54) | 2.38 (0.55)
Statistical Analysis 1: Comparison: Feedback Group vs Control Group; Test type: Superiority; p = 0.165, t-test, 2 sided; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [-0.45 to 2.64], Standard Error of Mean 0.79

2. Secondary Outcome: Change From Baseline in PROMIS Sleep T-score at 3-Month Follow up
Description: The 4-item PROMIS subscale for sleep was administered to participants at baseline and at 3 month follow up. The sleep subscale measures the extent to which patients experience problems with sleep over the past 7 days using a 5-point Likert scale. Higher scores reflect more severe sleep problems. To assess the effects of feedback on sleep, group differences in the change in PROMIS sleep T-scores from baseline to 3 month follow up (baseline PROMIS sleep T-score - 3 month PROMIS sleep T-score) were calculated. Positive change scores are indicative of improvement in sleep.
Time Frame: baseline and 3 month follow up
Population: Multiple imputation was used to determine follow-up scores for nonrespondents.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 151 | 149
T-score | 4.88 (0.76) | 4.04 (0.76)
Statistical Analysis 1: Comparison: Feedback Group vs Control Group; Test type: Superiority; p = 0.425, t-test, 2 sided; Mean Difference (Final Values) = 0.84, 95% CI 2-sided [-1.23 to 2.91], Standard Error of Mean 1.05

3. Secondary Outcome: Change From Baseline in PROMIS Pain T-score at 3-Month Follow up
Description: The 4-item PROMIS subscale for pain was administered to participants at baseline and at 3 month follow up. The pain subscale measures the extent to which patients experience problems with pain over the past 7 days using a 5-point Likert scale. Higher scores reflect greater pain. To assess the effects of feedback on pain, group differences in the change in PROMIS pain T-scores from baseline to 3-month follow up (baseline PROMIS pain T-score - 3 month PROMIS pain T-score) were calculated. Positive change scores are indicative of improvement in pain.
Time Frame: baseline and 3 month follow up
Population: Multiple imputation was used to determine follow-up scores for nonrespondents.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 151 | 149
T-score | 2.77 (0.68) | 2.12 (0.78)
Statistical Analysis 1: Comparison: Feedback Group vs Control Group; Test type: Superiority; p = 0.539, t-test, 2 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-1.41 to 2.70], Standard Error of Mean 1.05

4. Secondary Outcome: Change From Baseline in PROMIS Anxiety T-score at 3-Month Follow up
Description: The 4-item PROMIS subscale for anxiety was administered to participants at baseline and at 3 month follow up. The anxiety subscale measures the extent to which patients experience anxiety symptoms over the past 7 days using a 5-point Likert scale. Higher scores reflect greater anxiety. To assess the effects of feedback on anxiety, group differences in the change in PROMIS anxiety T-scores from baseline to 3-month follow up (baseline PROMIS anxiety T-score - 3 month PROMIS anxiety T-score) were calculated. Positive change scores are indicative of improvement in anxiety.
Time Frame: baseline and 3 month follow up
Population: Multiple imputation was used to determine follow-up scores for nonrespondents.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 151 | 149
T-score | 2.96 (0.77) | 2.13 (0.84)
Statistical Analysis 1: Comparison: Feedback Group vs Control Group; Test type: Superiority; p = 0.471, t-test, 2 sided; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-1.44 to 3.11], Standard Error of Mean 1.16

5. Secondary Outcome: Change From Baseline in PROMIS Depression T-score at 3-Month Follow up
Description: The 4-item PROMIS subscale for depression was administered to participants at baseline and at 3 month follow up. The depression subscale measures the extent to which patients experience depressive symptoms over the past 7 days using a 5-point Likert scale. Higher scores reflect greater depression. To assess the effects of feedback on depression, group differences in the change in PROMIS depression T-scores from baseline to 3-month follow up (baseline PROMIS depression T-score - 3 month PROMIS depression T-score) were calculated. Positive change scores are indicative of improvement in depression.
Time Frame: baseline and 3 month follow up
Population: Multiple imputation was used to determine follow-up scores for nonrespondents.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 151 | 149
T-score | 3.08 (0.77) | 1.59 (0.77)
Statistical Analysis 1: Comparison: Feedback Group vs Control Group; Test type: Superiority; p = 0.174, t-test, 2 sided; Mean Difference (Final Values) = 1.49, 95% CI 2-sided [-0.66 to 3.65], Standard Error of Mean 1.10

6. Secondary Outcome: Change From Baseline in PROMIS Fatigue T-score at 3-Month Follow up
Description: The 4-item PROMIS subscale for fatigue was administered to participants at baseline and at 3 month follow up. The fatigue subscale measures the extent to which patients experience problems with fatigue over the past 7 days using a 5-point Likert scale. Higher scores reflect greater fatigue. To assess the effects of feedback on fatigue, group differences in the change in PROMIS fatigue T-scores from baseline to 3-month follow up (baseline PROMIS fatigue T-score - 3 month PROMIS fatigue T-score) were calculated. Positive change scores are indicative of improvement in fatigue.
Time Frame: baseline and 3 month follow up
Population: Multiple imputation was used to determine follow-up scores for nonrespondents.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 151 | 149
T-score | 3.68 (0.87) | 2.01 (0.99)
Statistical Analysis 1: Comparison: Feedback Group vs Control Group; Test type: Superiority; p = 0.222, t-test, 2 sided; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [-1.00 to 4.35], Standard Error of Mean 1.36

7. Secondary Outcome: Treatment Satisfaction at 3-Month Follow-up
Description: At 3-month follow-up, treatment satisfaction was assessed. This 1-item measure assesses patients' satisfaction with the care of their symptoms overall on a 5-point Likert scale ranging from excellent to poor. Higher scores indicate poorer satisfaction.
Time Frame: 3 month follow-up
Population: Participants who responded to the treatment satisfaction question at 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Feedback Group | Control Group
Number analyzed (Participants) | 128 | 128
Participants
  Excellent | 25 | 21
  Very Good | 28 | 33
  Good | 39 | 42
  Fair | 22 | 26
  Poor | 14 | 6

8. Secondary Outcome: Sleep at 3-month Follow up, as Measured by the Pittsburgh Insomnia Rating Scale (PIRS-2)
Description: For this secondary outcome, data were collected from the group as a whole without regard to randomization. Thus, data is analyzed for the group as a whole rather than separately for each arm. At 3-month follow up, sleep was assessed using the 2-item Pittsburgh Insomnia Rating Scale (PIRS-2). PIRS-2 measures quality and satisfaction with sleep over the past week. Possible scores range from 0 to 6, with higher scores reflecting poorer sleep.
Time Frame: 3-month follow-up
Population: Participants who completed the PIRS-2 at 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Follow up Sample Responding to PIRS-2 (N=255): Of the 300 participants invited to complete the 3-month follow up assessment, 255 participants responded to items on the PIRS-2. No group comparisons were made.
Arm/Group | Follow up Sample Responding to PIRS-2 (N=255)
Number analyzed (Participants) | 255
units on a scale | 3.46 (1.80)

9. Secondary Outcome: Pain at 3 Month Follow up, as Measured by PEG
Description: For this secondary outcome, data were collected from the group as a whole without regard to randomization. Thus, data is analyzed for the group as a whole rather than separately for each arm. At 3-month follow up, pain was assessed using the 3-item PEG (Pain intensity, Enjoyment of life, and General activity). PEG measures pain intensity and interference in the past week. Possible scores range from 0 to 10, with higher scores reflecting more intense pain and interference.
Time Frame: 3 month follow up
Population: Participants who completed the PEG at 3 month follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Follow up Sample Responding to PEG (n=255): Of the 300 participants invited to complete the 3-month follow up assessment, 255 participants responded to items on PEG. No group comparisons were made.
Arm/Group | Follow up Sample Responding to PEG (n=255)
Number analyzed (Participants) | 255
units on a scale | 5.13 (3.28)

10. Secondary Outcome: Anxiety at 3 Month Follow up, as Measured by the Generalized Anxiety Disorder Scale (GAD-2)
Description: For this secondary outcome, data were collected from the group as a whole without regard to randomization. Thus, data is analyzed for the group as a whole rather than separately for each arm. At 3-month follow up, anxiety was assessed using the 2-item Generalized Anxiety Disorder scale (GAD-2). GAD-2 measures the frequency of anxiety symptoms over the past 2 weeks. Possible scores range from 0 to 6, with higher scores reflecting more severe anxiety.
Time Frame: 3 month follow up
Population: Participants who completed the GAD-2 at 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Follow up Sample Responding to GAD-2 (n=256): Of the 300 participants invited to complete the 3-month follow up assessment, 256 participants responded to items on the GAD-2. No group comparisons were made.
Arm/Group | Follow up Sample Responding to GAD-2 (n=256)
Number analyzed (Participants) | 256
units on a scale | 2.14 (2.08)

11. Secondary Outcome: Depression at 3-month Follow up, as Measured by the Patient Health Questionnaire (PHQ-2)
Description: For this secondary outcome, data were collected from the group as a whole without regard to randomization. Thus, data is analyzed for the group as a whole rather than separately for each arm. At 3-month follow up, depression was assessed using the 2-item Patient Health Questionnaire (PHQ-2). The PHQ-2 measures the frequency of depressive symptoms over the last 2 weeks. Possible scores range from 0 to 6, with higher scores reflecting more severe depression.
Time Frame: 3 month follow up
Population: Participants who completed the PHQ-2 at 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Follow up Sample Responding to PHQ-2 (n=255): Of the 300 participants invited to complete the 3-month follow up assessment, 255 participants responded to items on the PHQ-2. No group comparisons were made.
Arm/Group | Follow up Sample Responding to PHQ-2 (n=255)
Number analyzed (Participants) | 255
units on a scale | 2.06 (1.96)

12. Secondary Outcome: Fatigue at 3-month Follow up, as Measured by the SF-36 Vitality Scale
Description: For this secondary outcome, data were collected from the group as a whole without regard to randomization. Thus, data is analyzed for the group as a whole rather than separately for each arm. At 3-month follow up, fatigue was assessed using the 4-item SF-36 (Short Form-36 Healthy Survey) vitality scale. The SF-36 vitality scale measures fatigue and energy over the past week. Possible scores range from 0 to 100, with lower scores reflecting greater fatigue.
Time Frame: 3 month follow up
Population: Participants who completed the SF-36 vitality scale at 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Follow up Sample Responding to SF-36 Vitality Scale (n=256): Of the 300 participants invited to complete the 3-month follow up assessment, 256 participants responded to items on the SF-36 vitality scale. No group comparisons were made.
Arm/Group | Follow up Sample Responding to SF-36 Vitality Scale (n=256)
Number analyzed (Participants) | 256
units on a scale | 41.16 (22.34)

13. Secondary Outcome: Percentage of Participants With Laboratory Tests Ordered for SPADE Symptoms at Baseline Clinic Visit
Description: Electronic medical records were reviewed to determine the number of laboratory tests ordered for SPADE symptoms at the baseline clinic visit. The percentage of participants in each group with 0 or 1≤ lab tests ordered for SPADE symptoms at baseline was calculated.
Time Frame: baseline
Population: Participants whose electronic medical record of the baseline clinic visit was available for review
Measure: Number; unit: percentage of participants
Groups:
- Feedback Group (EMR): Patients whose clinician received baseline PROMIS symptom scores at the time of their clinic visit, and whose electronic medical record of the baseline clinic visit was available for review
- Control Group (EMR): Patients whose clinician did not receive baseline PROMIS symptom scores at the time of their clinic visit, and whose electronic medical record of the baseline clinic visit was available for review
Arm/Group | Feedback Group (EMR) | Control Group (EMR)
Number analyzed (Participants) | 147 | 145
percentage of participants
  Percentage of patients with 0 labs ordered | 91.8 | 90.3
  Percentage of patients with 1≤ labs ordered | 8.2 | 9.7

14. Secondary Outcome: Percentage of Participants With Radiologic (RAD) Tests Ordered for SPADE Symptoms at Baseline Clinic Visit
Description: Electronic medical records were reviewed to determine the number of radiologic (RAD) tests ordered for SPADE symptoms at the baseline clinic visit. The percentage of participants in each group with 0 or 1≤ RAD tests ordered for SPADE symptoms at baseline was calculated.
Time Frame: baseline
Population: Participants whose electronic medical record of the baseline clinic visit was available for review
Measure: Number; unit: percentage of participants
Arm/Group | Feedback Group (EMR) | Control Group (EMR)
Number analyzed (Participants) | 147 | 145
percentage of participants
  Percentage of patients with 0 RAD tests ordered | 86.4 | 84.1
  Percentage of patients with 1≤ RAD tests ordered | 13.6 | 15.9

15. Secondary Outcome: Percentage of Participants With Tests Ordered (Other Than Radiologic and Laboratory Tests) for SPADE Symptoms at Baseline Clinic Visit
Description: Electronic medical records were reviewed to determine the number of tests ordered, other than radiologic or laboratory tests (e.g., sleep study), for SPADE symptoms at the baseline clinic visit. The percentage of participants in each group with 0 or 1≤ tests ordered for SPADE symptoms at baseline was calculated.
Time Frame: baseline
Population: Participants whose electronic medical record of the baseline clinic visit was available for review
Measure: Number; unit: percentage of participants
Arm/Group | Feedback Group (EMR) | Control Group (EMR)
Number analyzed (Participants) | 147 | 145
percentage of participants
  Percentage of patients with 0 tests ordered | 91.2 | 97.9
  Percentage of patients with 1≤ tests ordered | 8.8 | 2.1

16. Secondary Outcome: Percentage of Participants With Medications Ordered for SPADE Symptoms at Baseline Clinic Visit
Description: Electronic medical records were reviewed to determine the number of medications ordered for SPADE symptoms at the baseline clinic visit. The percentage of participants in each group with 0, 1, 2, or 3≤ medications ordered for SPADE symptoms at baseline was calculated.
Time Frame: baseline
Population: Participants whose electronic medical record of the baseline clinic visit was available for review
Measure: Number; unit: percentage of participants
Arm/Group | Feedback Group (EMR) | Control Group (EMR)
Number analyzed (Participants) | 147 | 145
percentage of participants
  Percentage of patients with 0 meds ordered | 38.1 | 30.3
  Percentage of patients with 1 med ordered | 27.2 | 35.2
  Percentage of patients with 2 meds ordered | 19.1 | 23.5
  Percentage of patients with 3≤ meds ordered | 15.6 | 11.0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 20 month-period of time (March 2015 to October 2016).
Description: The definitions do not differ.
Arm/Group | Feedback Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/149
Other Adverse Events (participants affected / at risk) | 0/151 | 0/149

LIMITATIONS AND CAVEATS:
A convenience sample was obtained from urban primary care clinics. Further studies in different primary care populations are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes